CLINICAL TRIAL: NCT04062773
Title: A Pilot Study to Evaluate the Effect of Time-Restricted Feeding on Blood Glucose, Insulin Sensitivity and Quality of Life
Brief Title: Time-Restricted Feeding on Glucose Homeostasis and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA HM-2019-012
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2; Time Restricted Feeding
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: 12 week parallel trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRF (Experimental): Eating restricted to between midday and 6pm.
  Interventions: Behavioral: TRF
- Normal timing of food intake. (Placebo Comparator): Eating between 8am and 11pm.
  Interventions: Behavioral: Normal timing of food intake

INTERVENTIONS:
Behavioral: TRF — time restricted feeding group
  Arms: TRF
Behavioral: Normal timing of food intake — no time restricted feeding
  Arms: Normal timing of food intake.

SUMMARY:
Background: Time-restricted feeding can improve insulin sensitivity, and increase fat oxidation in people with prediabetes independent of weight loss. It may also help people to lose weight. However, it has not been tested in people with type 2 diabetes.

Plan of investigation: Participants meeting the eligibility criteria will be randomized to the TRF arm or the continuous eating arm. Both arms with be given a prescribed dietary plan to help them lose 5% of body weight. In the TRF they will permitted to eat between midday and 6pm. In the continuous eating arm they will be allowed to eat between 8am and 11pm. Participants will attend the nutrition clinic every two weeks to be weighed and be given personalized support to help them follow their assigned diet. Prior to starting the diets outcome measures will be taken: Glycaemia will be measured by a glucose tolerance test, and 7-day continuous glucose monitoring. HbA1c will be taken from fasting blood sample. In addition, the fasting sample will be taken for measurement of insulin, lipid profile and inflammatory markers. We will also use questionnaires to assess quality of life, a 3-day food diary to assess compliance to diet especially meal timings. Capillary ketones will also be used to assess whether compliance to the assigned fasting period. Outcome measures will also be taken during 7 days of the second month, and then the final seven days of the last month on the diet. The primary outcome is HbA1c.

DETAILED DESCRIPTION:
Experimental Design

12-week parallel randomised control trial

Recruitment

We will recruit via advertisements outside Dasman using social media and local ads in addition to screening of Dasman Registry for any potential participants. Opportunistic recruitment will also occur by DDI dietitians. Following telephone screening to ensure the potential participant meets initial screening criteria we will carry out a medical screening to ensure the person can take part.

Environment All screening, dietary counselling visits, and placement of the CGM will take place at the Dasman Diabetes Institute (DDI). The institute has extensive space for interventional studies, including screening rooms, body composition assessment and clinical rooms for placement of the CGM monitor.

STUDY INTERVENTIONS

For both groups all participants will be guided towards a 5% weight loss based on individualised energy requirements. The difference will be the hours during which the participants consume their required calories.

* Time restricted feeding group: Will consume their calories between 12pm and 6pm.
* Continuous energy restriction group: Will consume their calories between 8am and 11pm.

Participants will be guided towards their weight loss during one-to-one visits at baseline and every 2 weeks for 12 weeks.

Procedures

* At baseline and follow-up all participants will undergo an oral glucose tolerance test.
* A blood sample will also be taken for HbA1c, lipid profile, fasting insulin, inflammatory factors and a sample for Biobank. The biobank sample will be stored to enable us, with other researchers at DDI to understand the heterogeneity of type 2 diabetes; whether certain people respond to dietary interventions based on their genetic, epigenetic or metabolomic background; and ultimately will help guide clinical care.
* Participants will wear Flash Glucose monitoring or other continuous glucose monitoring device to measure their 24-hour blood glucose concentrations during the seven days preceding the start of the dietary intervention, seven days of the second month, and the final seven days of the third month.
* Participants will also measure their capillary ketones during the first three days of the first month, three days of the second month, and final three days of the third month.
* Medication changes: prandial medications (insulin or sulphonylurea) will be altered to the timing of meal intake. Any reduction in medication due to changes in glucose will be carried out by the patient's doctor.
* A quality of life questionnaire: PAID.
* A 3 day food diary with meal times to check compliance.

Statistical Methods

This is a pilot study. We will recruit 25 people per group. This is based on recommendations for sample sizes for feasibility and pilot studies.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to follow time restricted feeding protocol if randomized to the TRF arm.
* Age 21-65 years
* T2DM with any diabetes medication
* BMI of 25-45 kg/m2
* Wake up at a regular time between 5-8 am
* Able to provide informed consent.

Exclusion Criteria:

* Weight loss of more than 5 kg within the past 6 months
* HbA1c of <6·5% and >12%
* Serious current or recent illness including cancer or severe or unstable heart failure.
* Participation in another clinical research trial.
* Current treatment with anti-obesity drugs.
* Substance abuse
* Learning difficulties
* Presence of an eating disorder
* Purging behaviour
* Pregnancy or consideration of pregnancy
* Hospital admission for depression or use of antipsychotic drugs.
* Regularly eat within a <9-hour period each day
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Change in HbA1c between the intervention and control arms.

SECONDARY OUTCOMES:
Body weight | 12 weeks
  Change in body weight between the intervention and control arms.
Insulin sensitivity | 12 weeks
  Change insulin sensitivitiy assessed by OGTT between the intervention and control arms.
Diabetes medications | 12 weeks
  Change in diabetes medications between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in TNF-alpha in pg/mL between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in IL-10 in pg/mL between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in IL-6 in pg/mL between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in IL-18 in pg/mL between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in CRP in mg/L between the intervention and control arms.
Inflammatory markers | 12 weeks
  Change in adiponectin in µg/mL the intervention and control arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait